CLINICAL TRIAL: NCT04064541
Title: Virtual Visits and Distance Health to Optimize Research Trial Offerings to Heart Failure Patients: An Innovative Approach
Brief Title: Virtual Visits to Optimize Research Trial Offerings to HF Patients
Acronym: Optimize-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Laurie Ann Moennich, Principal Investigator, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-818
Record Dates: First submitted 2019-08-02; First posted 2019-08-22 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Heart Failure, Systolic; Heart Failure With Preserved Ejection Fraction
Keywords: Heart Failure; Distance Health; Virtual Visits; Functional Assessment; Quality of Life; Cognitive Assessment
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure

STUDY DESIGN:
Intervention Model Description: Subjects in this study will serve as their own control in order to assess their ability to perform functional, cognitive and QOL assessments in the virtual/ distance health environment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Visit (Other): At the baseline visit patients will complete an in-clinic baseline visit consisting of Medical Hx review, NYHA assessment, Questionnaires (EQ-5D-5L, KCCQ, Frailty Index for Elders & Mini Cog) and Functional Assessments (Timed Up & Go and 6MWT). Patients will also receive virtual visit training and complete an in-clinic virtual visit consisting of the previously stated functional assessments.
  All follow-up visits will occur via virtual distance health visits. These f/u visits will occur at Day 7and Day 14 At the initiation of each distance health f/u visit the patient's current state of health will be assessed as well as NYHA. Patient Questionnaires(EQ-5D-5L, KCCQ & Frailty Index) and Functional Assessments(Timed Up & Go and 6MWT) will be completed.
  Interventions: Other: Virtual Visit

INTERVENTIONS:
Other: Virtual Visit — Virtual Visit

SUMMARY:
This pilot study seeks to understand if distance health technology with virtual visits hold the key to improving access for patients who wish to partake in clinical trials clearing barriers to enrollment.

DETAILED DESCRIPTION:
Patient participation in clinical trials is crucial to ultimately shaping change in care delivery and development of new treatments that improve quality of life and meaningful patient outcomes. While they hold much value, the time and resources patients must allot to participation in protocol requirements of some clinical trials can be a barrier to trial enrollment. With the advent of Distance Health, and Virtual Visits in particular, accompanied by an increase in patient utilization of home computers and smart phones, patients are swarming to different communication platforms with their care providers. We hypothesize that distance health technology with virtual visits hold the key to improving access for patients who wish to partake in clinical trials, clearing barriers to enrollment.

If the virtual administration of clinical trial assessments is non-inferior to the tests regularly administered during in-clinic research related visits, this approach should be adopted by industry-sponsored and investigator initiated research studies in heart failure cohorts. If patients have the technological means and willingness to participate in the study, the ability to perform these tests in the comfort of their own home will likely make clinical trial enrollment more attractive and feasible for the patient. Furthermore, increasing clinical trial enrollment by diminishing access barriers will improve patient care by including a more diverse patient population in study enrollment and decrease study follow up attrition rates.

At the baseline visit prior to consent, potential subjects will be shown the distance of 30-50 feet while in the clinic setting, in order to determine if walking distance is feasible in the home environment. Once consented patients will complete an in-clinic baseline visit consisting of Medical Hx review, New York Hospital Association (NYHA) assessment, Questionnaires (EQ-5D-5L, KCCQ, Frailty Index for Elders & Mini Cog) and Functional Assessments (Timed Up & Go and 6MWT). Patients will also receive virtual visit training. Efforts will be made to enroll subjects from all the various NYHA class distinctions (II,III,IV). A baseline virtual visit will be completed in the clinic setting to ensure patient can perform the functional portion of the virtual visit in the home.

All follow-up visits will occur via virtual distance health visits. These f/u visits will occur 2 times after the initial baseline visit (Day 7and Day 14 [+/- 3 days for all f/u time points]. It is felt that 2 f/u visits completed in the home will reflect adequate data regarding feasibility for performing the procedures in the home environment while also reflecting the real time changing functional fluctuations of the patient with chronic HF. At the initiation of each distance health f/u visit the patient's current state of health will be assessed as well as NYHA. Questions will be asked of the patient to assess any changes in medical condition since the previous visit. Visit procedures will be rescheduled if the patient indicates that they are not feeling up to completing the study procedures on the scheduled day. Patient Questionnaires(EQ-5D-5L, KCCQ & Frailty Index) and Functional Assessments(Timed Up & Go and 6MWT) will be completed.

In order to complete the study procedures in the home during the distance health visits, patients will be provided with 2 cones and a measuring tape for marking the distances for the functional assessment tests.

If at anytime, the subject indicates distress or injury (ex: falling) while performing study procedures, the research staff will call 911 on the patient's behalf.

ELIGIBILITY:
Inclusion Criteria:

1. Males or Females
2. Aged >18 years
3. Diagnosed with HFpEF (preserved EF) or HFrEF (reduced EF)
4. Patient has a distance to walk at home of at least 10m/30 feet up to a maximum 15m/50 feet.

   The distance anticipated to be used at home is to be used in clinic)(Ex: 1-3 average car lengths, width of a high school basketball court, 2/3 to1and2/3 lengths of a tour bus, 30-50 rulers end to end, 30-50 sub-sandwiches end to end)
5. Having standard of care clinical evaluations performed at the Cleveland Clinic Main Campus.
6. Willing to perform distance health evaluations during study participation.
7. Patient or an individual in their social support network has the equipment (phone, computer, tablet) and internet connection to perform a distance health research visit.

Exclusion Criteria:

1. Unstable Angina or Myocardial infarction within the past 1 month.
2. History of Heart Transplant or actively listed for heart or any solid organ or tissue transplant
3. Implanted with an left ventricular assist device (LVAD)
4. Scheduled to be implanted with a left ventricular assist device (LVAD) within 45 days of signing consent.
5. Currently residing at a nursing home or rehabilitation facility.
6. Currently receiving Hospice services
7. Malignancy or other condition limiting life expectancy to less than 6 months.
8. Inability to walk without assist (cane is acceptable)
9. Inability or unwillingness to comply with study requirements in the opinion of the investigator
10. Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Patient's ability to complete the American Thoracic Society 6-minute walk test functional assessment via a virtual visit at Day 7 as compared to completing the same baseline test in the outpatient clinic. | Day 7
  Patients will perform the American Thoracic Society 6-minute walk test (6MWT) per a virtual visit initially in the outpatient clinical area and then from their home environment. The visit performed in the outpatient clinical area will be the baseline data.The distance of each lap walked will range from 30-50 feet. The patients will be timed for 6 minutes and laps counted by the study coordinator via the virtual visit. Pre and post test, the patient will be asked to rate their dyspnea and fatigue as per the Borg Scale. The dyspnea & fatigue Borg Scale ranges will be from 0 (no distress) to 11 (maximum distress). The results of the distance walked and fatigue and dyspnea scales will be evaluated at each visit time point to determine the reliability & validity of the patient's ability to successfully perform the test via a virtual visit. The patient will be their own control.
Patient's ability to complete the American Thoracic Society 6-minute walk test functional assessment via a virtual visit at Day 14 as compared to completing the same baseline test in the outpatient clinic. | Day 14
  Patients will perform the American Thoracic Society 6-minute walk test (6MWT) per a virtual visit initially in the outpatient clinical area and then from their home environment. The visit performed in the outpatient clinical area will be the baseline data.The distance of each lap walked will range from 30-50 feet. The patients will be timed for 6 minutes and laps counted by the study coordinator via the virtual visit. Pre and post test, the patient will be asked to rate their dyspnea and fatigue as per the Borg Scale. The dyspnea & fatigue Borg Scale ranges will be from 0 (no distress) to 11 (maximum distress). The results of the distance walked and fatigue and dyspnea scales will be evaluated at each visit time point to determine the reliability & validity of the patient's ability to successfully perform the test via a virtual visit. The patient will be their own control.
Patient's ability to complete the Timed Up and Go functional assessment test via virtual visit at Day 7 as compared to completing the same baseline test in the outpatient clinic. | Day 7
  Patients will perform the Timed Up and Go functional assessment test per a virtual visit initially in the outpatient clinical area and then from their home environment. Patients will complete 2-10 foot laps. The patients will be observed (posture), timed and laps counted by the study coordinator via the virtual visit. Data collected at each time point will be will be used to determine the reliability and validity of conducting this test as a virtual visit in the home environment. The patient will be their own control
Patient's ability to complete the Timed Up and Go functional assessment test via virtual visit at Day 14 as compared to completing the same baseline test in the outpatient clinic. | Day 14
  Patients will perform the Timed Up and Go functional assessment test per a virtual visit initially in the outpatient clinical area and then from their home environment. Patients will complete 2-10 foot laps. The patients will be observed (posture), timed and laps counted by the study coordinator via the virtual visit. Data collected at each time point will be will be used to determine the reliability and validity of conducting this test as a virtual visit in the home environment. The patient will be their own control
Patient's ability to complete the Kansas City Cardiomyopathy Quality of Life Questionnaire (KCCQ) per virtual visit at Day 7 as compared to completing the same baseline test in the outpatient clinic. | Day 7
  Kansas City Cardiomyopathy Questionnaire assesses heart failure effects on life over the past 2 weeks. 8 sections, 12 questions. #1-Activity. Response range- Extremely Limited= 1 to of Not limited for other reasons or did not do the activity= 6. #2-Swelling. Response range- Every morning =1 to Never= 5. #3/ #4 -Fatigue and Shortness of breath. Response range-All of the time = 1 to Never =7. #5-Shortness of breath/Sleep. Response range-Every night= 1 to Never= 5. #6-Enjoyment of life. Response range-Extremely limited= 1 to Not limited at all=5. #7 -Perception of life. Response range-Not at all satisfied= 1 to Completely satisfied= 5. #8-Lifestyle. Response range-Severely limited=1 to Does not apply or did not do for other reasons = 6. Overall questionnaire total score range-12 to 70 points. The higher the score the less impact heart failure has on quality of life.
Patient's ability to complete the Kansas City Cardiomyopathy Quality of Life Questionnaire (KCCQ) per virtual visit at Day 14 as compared to completing the same baseline test in the outpatient clinic. | Day 14
  Kansas City Cardiomyopathy Questionnaire assesses heart failure effects on life over the past 2 weeks. 8 sections, 12 questions. #1-Activity. Response range- Extremely Limited= 1 to of Not limited for other reasons or did not do the activity= 6. #2-Swelling. Response range- Every morning =1 to Never= 5. #3/ #4 -Fatigue and Shortness of breath. Response range-All of the time = 1 to Never =7. #5-Shortness of breath/Sleep. Response range-Every night= 1 to Never= 5. #6-Enjoyment of life. Response range-Extremely limited= 1 to Not limited at all=5. #7 -Perception of life. Response range-Not at all satisfied= 1 to Completely satisfied= 5. #8-Lifestyle. Response range-Severely limited=1 to Does not apply or did not do for other reasons = 6. Overall questionnaire total score range-12 to 70 points. The higher the score the less impact heart failure has on quality of life.
Patient's ability to complete the Frailty Index for Elders (FIFE) questionnaire per virtual visit at Day 7 as compared to completing the same baseline test in the outpatient clinic. | Day 7
  The Frailty Index for Elders (FIFE) assesses for frailty risk in older adults. The risk for becoming frail increases as older adults live longer with chronic illnesses. Frailty is a geriatric syndrome affecting older adults due to multisystem decline that increases vulnerability to poor health effects. FIFE is a 10-item assessment instrument with responses of yes=1 to No=0.Scores range from 0-10. A score of 0 indicates no frailty; a score of 1-3 indicates frailty risk; and a score of 4 or greater indicates frailty. Questions include patient's perception of activity, self- care, weight changes, tooth/mouth issues, appetite, social activities, overall health, fatigue, hospitalization within past 3 months and emergency room visits over past 3 months. Data will be used to determine reliability and validity to complete this questionnaire as a virtual visit.
Patient's ability to complete the Frailty Index for Elders (FIFE) questionnaire per virtual visit at Day 14 as compared to completing the same baseline test in the outpatient clinic. | Day 14
  The Frailty Index for Elders (FIFE) assesses for frailty risk in older adults. The risk for becoming frail increases as older adults live longer with chronic illnesses. Frailty is a geriatric syndrome affecting older adults due to multisystem decline that increases vulnerability to poor health effects. FIFE is a 10-item assessment instrument with responses of yes=1 to No=0.Scores range from 0-10. A score of 0 indicates no frailty; a score of 1-3 indicates frailty risk; and a score of 4 or greater indicates frailty. Questions include patient's perception of activity, self- care, weight changes, tooth/mouth issues, appetite, social activities, overall health, fatigue, hospitalization within past 3 months and emergency room visits over past 3 months.
Patient's ability to complete the European Quality Of Life-5Dimension-5Level (EQ-5D-5L) Health State Questionnaire per virtual visit at Day 7 as compared to completing the same baseline test in the outpatient clinic. | Day 7
  European Quality Of Life-5Dimension-5Level has 2 sections: 1) health state & 2) evaluation. 1) measures health state using 5 dimensions -limitations in mobility/self-care/usual activities/pain or discomfort & anxiety or depression. Each dimension has 5 response levels -1=no problems/2=slight problems/3=moderate problems/4=severe problems & 5=unable to do/having extreme problems. A level from each dimension defines health state. States are expressed as 5 digit codes. Ex: state 11111= no problems on any of the 5 dimensions, while state 12345= no problems mobility, slight problems washing or dressing, moderate problems doing usual activities, severe pain or discomfort & extreme anxiety or depression. 2) evaluates overall health status using European Quality of Life Visual Analog Scale. "X" is marked on a vertical scale with end points of 0 =worst health you can imagine and 100=best health you can imagine. Number marked=quantitative measure of health
Patient's ability to complete the European Quality Of Life-5Dimension-5Level (EQ-5D-5L) Health State Questionnaire per virtual visit at Day 14 as compared to completing the same baseline test in the outpatient clinic. | Day 14
  European Quality Of Life-5Dimension-5Level has 2 sections: 1) health state & 2) evaluation. 1) measures health state using 5 dimensions -limitations in mobility/self-care/usual activities/pain or discomfort & anxiety or depression. Each dimension has 5 response levels -1=no problems/2=slight problems/3=moderate problems/4=severe problems & 5=unable to do/having extreme problems. A level from each dimension defines health state. States are expressed as 5 digit codes. Ex: state 11111= no problems on any of the 5 dimensions, while state 12345= no problems mobility, slight problems washing or dressing, moderate problems doing usual activities, severe pain or discomfort & extreme anxiety or depression. 2) evaluates overall health status using European Quality of Life Visual Analog Scale. "X" is marked on a vertical scale with end points of 0 =worst health you can imagine and 100=best health you can imagine. Number marked=quantitative measure of health

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Ann Moennich, MPH CPH, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No